CLINICAL TRIAL: NCT00396968
Title: AMD3100 With Busulfan, Fludarabine and Thymoglobulin for Allogeneic Stem Cell Transplantation for Acute Myelogenous Leukemia and Myelodysplastic Syndromes
Brief Title: AMD3100 With Busulfan, Fludarabine and Thymoglobulin for Allogeneic Stem Cell Transplant for AML and MDS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: AnorMED (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-2201
Record Dates: First submitted 2006-11-06; First posted 2006-11-08 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes
Keywords: AMD3100; Acute Myelogenous Leukemai; Myelodysplastic Syndromes; Allogeneic stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — plerixafor

INTERVENTIONS:
Drug: AMD3100
Procedure: Allogeneic Stem Cell Transplantation

SUMMARY:
AMD3100 given in combination with busulfan, fludarabine (and thymoglobulin (ATG) for unrelated or HLA nonidentical donors) preparative regimen in patients with acute myelogenous leukemia (AML) / myelodysplastic syndromes (MDS).

This study aims to determine if in AML and MDS patients there is a reduction of malignant cells and enhanced elimination of the leukemia as assessed by progression free survival. Secondary goals will be to assess effects on engraftment, graft versus host disease (GVHD) and immune reconstitution.

DETAILED DESCRIPTION:
This is a single centre phase I/II study which will be conducted in two stages. The ability of AMD3100 to augment the antileukemic effect of chemotherapy and stem cell transplantation in patients with MDS or with AML in first or subsequent relapse, second or greater remission or primary induction failure will be assessed.

The primary objective in Stage 1 is to determine an acceptably safe dose, utilizing the continual reassessment method (CRM).The CRM is a model-based statistical procedure for conducting phase I clinical trials that assigns doses to successive cohorts of patients based on the doses given and outcomes observed (toxicity or no toxicity) of all previous patients. In this sense, the method is "outcome-adaptive." The CRM relies on a simple Bayesian model for the probability of toxicity as a function of dose. As the dose-toxicity data in the trial accumulate the Bayesian model "learns" about the relationship between dose and probability of toxicity. Numerous computer simulation studies (and the references therein) have shown that the CRM has greatly superior properties compared to conventional "3+3" algorithms. This is due to the facts that conventional algorithms are not model-based, they only use data from the most recent 6 patients, and they tend to stop the trial very early, with the consequences that they are very likely to give very unreliable estimates of the toxicity probability at each dose and provide an unreliable recommended maximum tolerated dose (MTD).

Under the particular version of the CRM being used in this trial, following treatment of the first cohort of three patients at the initial dose level 80 µg/kg, the following decisions are possible:

* If 0 of the first 3 patients (#1, 2 and 3) experience toxicity, then the method will escalate and the second cohort of patients (#4, 5 and 6) will be treated at the second dose level, 160 µg/kg.
* If either 1 or 2 of the first 3 patients experience toxicity, then the method will stay at the starting dose, so the second cohort will be treated at the lowest dose level, 80 µg/kg.
* If all 3 of the first 3 patients experience toxicity, then the posterior probability that the lowest dose is unacceptably toxic will be 0.951, and since this exceeds the decision cut-off 0.90 in the protocol the phase I trial will be terminated with the conclusion that the lowest dose level 80 µg/kg is excessively toxic.

If the trial continues, for all successive cohorts after the first, since the decision of which dose to assign utilizes all of the dose-toxicity data from all patients treated previously, there are too many possibilities to enumerate. For example, there are 12 possible outcomes for the second cohort, and this number increases exponentially as the trial progresses. However, at any point in the trial, the estimated probability of toxicity at each dose based on the most recent data may easily be estimated and this information made available to the investigators. Additional safety provisions are that the middle dose of 160 µg/kg may not be skipped when initially escalating from 80 µg/kg, and the trial will be terminated early with no dose chosen if the lowest dose is excessively toxic.

The primary objective in Stage 2 is to determine progression free survival post-allogeneic transplant, in terms of time to treatment failure and survival. Stage 1 will include both prognostic subgroups CR and not in complete remission (NCR). In Stage 2, different monitoring rules will be used in CR and NCR subgroups to reflect their very different historical failure rates. Additionally, all patients treated at the dose selected in Stage 1 will be counted as members of the Stage 2 sample.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML past first remission, (i.e., in first or subsequent relapse, in second or greater remission or primary induction failure) or MDS with intermediate or high risk International Prognostic Scoring System (IPSS) score (71) or having failed to respond or recurred after chemotherapy.
* WBC <20 x 10e9/l.
* Patients should have a histocompatible, related or unrelated volunteer donor available for a PBSC transplant. A histocompatible donor is defined as HLA matched for at least 9 of 10 HLA A, B, C, DR and DQ antigens by high-resolution DNA technique per departmental routine.
* Patient has not been administered any other systemic chemotherapeutic drug (including Mylotarg) within 21 days prior to trial enrollment. (Hydroxyurea is permitted if indicated to control induction refractory disease, and intrathecal (IT) chemotherapy is allowed if indicated as maintenance treatment for previously diagnosed leptomeningeal disease (LMD), that has been in remission for at least 3 months prior to enrollment on this study).
* Zubrod performance status < 2.
* Left ventricular ejection fraction >45%. No uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease. This should be performed within 28 days prior to study entry.
* No symptomatic pulmonary disease. Forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC) and diffusion capacity of carbon monoxide (DLCO) > 50 % of expected, corrected for hemoglobin. This should be performed within 28 days prior to study entry.
* Serum creatinine <1.5 mg/dl.
* Serum glutamic pyruvic transaminase (SGPT) <200 IU/ml. Total serum bilirubin and alkaline phosphatase <2.5 times laboratory standard upper limit of normal (ULN), or considered not clinically significant by the protocol PI.
* Patient or patient's legal representative able to sign informed consent.

Exclusion Criteria:

* HIV positive.
* Female patient who is pregnant (negative pregnancy test is required for all women of child-bearing-potential).
* Pleural/pericardial effusion or ascites estimated > 1 liter.
* Uncontrolled infection. Patients considered to have uncontrolled infections including active fungal pneumonia are not eligible. Patients with infections or pulmonary infiltrates responding to antimicrobial treatment are eligible. Infectious Disease consultation should be obtained if indicated. These cases should be discussed with the Protocol PI who is the final arbiter of eligibility.
* Evidence of chronic active hepatitis or cirrhosis.
* Patients should not have received investigational agent(s) or intensive chemotherapy within 21 days of starting the study treatment regimen.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
To determine if AMD3100 given in a sequential dose escalation at 80, 160 and 240 µg/kg in combination with busulfan, fludarabine (and ATG for unrelated or HLA nonidentical donors) for treatment of AML/MDS:
Stage 1 - Is Safe
Stage 2 - Will improve progression free survival post allogeneic stem cell transplantation from an HLA compatible donor compared to historical controls.

SECONDARY OUTCOMES:
Stage 2 - Determine the time from stem cell transplant to PMN engraftment compared to historical controls.
Determine the rate and severity grading of GVHD compared to historical controls.
Determine immune reconstitution compared to historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company